CLINICAL TRIAL: NCT03238144
Title: Tissue Stresses of Cancer: A Phase I/II,Multi-centre, Feasibility Study to Image the Tissue Stiffness/Stresses to Predict Outcome in Breast Cancer
Brief Title: Tissue Stresses of Cancer (Force Horizon 2020)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 204546
Record Dates: First submitted 2016-11-24; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRF +/-contrast enhanced MRI (Other): MRF with or without contrast enhanced MRI
  Interventions: Other: MRF scan

INTERVENTIONS:
Other: MRF scan — MRF with or without dynamic contrast-enhanced MRI scans.

SUMMARY:
This project is investigating a novel MRI method called Magnetic Resonance Force (MRF). MRF has been developed to accurately estimate tumour stiffness in the breast by measuring the interstitial fluid pressure (IFP).

50 healthy volunteers will be recruited to extend the hardware and establish MRF imaging acquisition protocols for pre and post-menopausal women. Once completed, we will test this new imaging technique with the acquired imaging protocols on 100 patients undergoing surgery as first line of their treatment for their breast cancer to establish a potential biomarker signature predictive of lymph node involvement and metastatic potential. Simultaneously, 50 patients undergoing chemotherapy as first line of their treatment for their breast cancers will be recruited to develop a biomarker signature that could predict response or resistance to neoadjuvant chemotherapy as determined by conventional imaging and histopathology.

DETAILED DESCRIPTION:
Magnetic Resonance Force (MRF) is based on Magnetic Resonance Elastography which uses mechanical waves to quantitatively assess the viscoelastic properties of tumours and the shift in interstitial fluid pressure (or stiffness) of tissues.

It generates 3D images of applied deformation via low frequency acoustic waves within the tissue and provides a snapshot of the apparent stiffening of the tumour border zone. Growth induced stretch of the tumour not only increases stiffness but also alters the apparent change in stiffness due to additional loading. Magnetic Resonance Force (MRF) provides measures of MRE and macro-deformation at multiple load states therefore enabling estimation of tissue properties as well as the stress load relation. Since the stress load relation is related to tumour swelling and modifications, it can be directly linked to the tumour pre-strain and provides an indicator of the underlying interstitial tumour pressure. Using biomechanical models it is possible to directly translate the stress load relation into an estimate of IFP. The same approach also allows quantifying the active pull by cell traction forces (CTFs) coming from the tumour and exerted onto its surroundings. While that force is directed inwards, the force generated by the elevated interstitial fluid pressure (IFP) is directed outwards allowing separation of both effects from each other. These forces represent one of the biomarkers which we will quantify within the this project using MRF.

ELIGIBILITY:
Inclusion Criteria for healthy Volunteers:

* Healthy female pre- and post-menopausal volunteers ≥ 40 years of age
* Pre-menopausal patients between the age of 40-55 years of age will have two scans:

  1. Between day 7- 15 of their menstrual cycle and
  2. Between day 21-28 of their menstrual cycle
* Postmenopausal patients of 55 years and above will have one scan only.
* No prior history of breast cancer
* Written informed consent to participate in this study

Inclusion Criteria for patients undergoing primary surgery:

* Females ≥ 18 years of age with a diagnosis of invasive breast cancer with tumour size of at least 5mm as determined by USS
* Scheduled to undergo breast conserving surgery or mastectomy +/- sentinel lymph node biopsy or axillary lymph node dissection
* Written informed consent to participate in this study.

Inclusion Criteria for patients undergoing neoadjuvant chemotherapy:

* Females ≥ 18 years of age with a diagnosis of invasive breast cancer
* Scheduled to undergo neoadjuvant systemic chemotherapy
* Written informed consent to participate in this study.

Exclusion Criteria for healthy volunteers:

Contraindications for MRI such as:

* cardiac pacemaker
* metallic implants
* major claustrophobia
* pregnancy or breastfeeding
* Inability to provide written informed consent

Exclusion Criteria for patient undergoing primary surgery and neoadjuvant chemotherapy:

* Contraindications for MRI such as:
* cardiac pacemaker
* metallic implants
* major claustrophobia
* prior breast cancer treatment
* pregnancy or breastfeeding
* known allergy against the contrast agent (gadolinium chelate) and renal failure
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of reduction in interstitial fluid pressure confirmed by MRF | up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St.Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sinha AP, Jurrius P, van Schelt AS, Darwish O, Shifa B, Annio G, Peterson Z, Jeffery H, Welsh K, Metafa A, Spence J, Kothari A, Hamed H, Bitsakou G, Karydakis V, Thorat M, Shaari E, Sever A, Rigg A, Ng T, Pinder S, Sinkus R, Purushotham A. Tumor Biomechanics Quantified Using MR Elastography to Predict Response to Neoadjuvant Chemotherapy in Individuals with Breast Cancer. Radiol Imaging Cancer. 2025 Mar;7(2):e240138. doi: 10.1148/rycan.240138. PMID 39950962